CLINICAL TRIAL: NCT05404139
Title: Duration of Androgen Receptor Pathway Inhibitor and ADT With Metastasis Directed Therapy in Oligometastatic Cancer of the Prostate
Brief Title: Duration of Androgen Receptor Pathway Inhibitor and ADT With Metastasis Directed Therapy in Oligometastatic Cancer of the Prostate (DIRECT)
Acronym: DIRECT
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22-5274
Record Dates: First submitted 2022-05-19; First posted 2022-06-03 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — enzalutamide; Androgen Antagonists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 - Standard of Care (Other): Participants in this group will receive standard of care radiation treatment and ADT. Participants will start ADT first. Androgen deprivation therapy will be delivered via injection every 4 months as per standard of care (for 8 months total). At the same time, or within 3 months of starting ADT, participants will begin radiation treatment. The radiation treatment course will consist of 2-5 sessions of radiation daily or every other day (the number of sessions will be determined by the physician depending on the location of cancer, number of cancer spots, etc.).
  Interventions: Other: Standard of Care SBRT and ADT
- Arm 3 - Study Treatment (Experimental): Participants in this group will receive standard of care radiation treatment and ADT, plus abiraterone. Participants will start ADT first. Androgen deprivation therapy will be delivered via injection every 4 months as per standard of care (for 8 months total). At the same time, or within 3 months of starting ADT, participants will begin radiation treatment. The radiation treatment course will consist of 2-5 sessions of radiation daily or every other day (the number of sessions will be determined by the physician depending on the location of cancer, number of cancer spots, etc.). In addition, participants will take abiraterone orally (by mouth) daily for 8-9 months. Participants will start the first pill within a month of enrollment. This pill can be taken around the same time of day with or without food.
  Interventions: Drug: Enzalutamide; Other: Standard of Care SBRT and ADT

INTERVENTIONS:
Drug: Enzalutamide — Second-generation androgen pathway inhibitor (ARAT), oral tablet
  Arms: Arm 3 - Study Treatment
Other: Standard of Care SBRT and ADT — Standard of care stereotactic body radiation therapy (SBRT) and androgen deprivation therapy (ADT)

SUMMARY:
This is a multi-centre, investigator-initiated, two-arm, randomized trial to investigate the addition on androgen receptor pathway inhibitor to standard of care radiation and hormone therapy improve quality of life.

Participants will either receive standard of care radiation and hormone (ADT) therapy (Arm 1) or standard of care radiation and hormone (ADT) therapy plus oral abiraterone for 8-9 months (Arm 3). Participants will be routinely follow-up in clinic or remotely for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Able to provide informed consent
3. Histologic diagnosis of prostate adenocarcinoma
4. ECOG performance status 0-2
5. Stage IV castrate sensitive metachronous metastatic prostate cancer. diagnosed within 6 months of study enrollment with 1-10 metastases

   1. Maximum one metastatic deposit on conventional imaging (CT or bone scan or MR)
   2. Additional metastases can be detectable by PSMA PET only
6. All sites of disease are amenable to and can be safely treated with radiotherapy
7. Patients decline continuous use of ADT

Exclusion Criteria:

1. Significant comorbidities rendering patient not suitable for ADT, enzalutamide and SBRT
2. History of malignancy within the past 5 years, excluding non-melanoma skin cancer and in-situ cancer, managed non-curatively
3. Prior use of salvage systemic therapy
4. Evidence of spinal cord compression

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male participants only as this study is in metastatic prostate cancer.
Enrollment: 132 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 5 years
  Determine if progression free survival improves with the addition of intermittent enzalutamide to standard of care treatment.

SECONDARY OUTCOMES:
Patient-reported quality of life | 5 years
  Determine if the addition of intermittent enzalutamide to standard of care treatment results in a patient-reported quality of life difference compared to standard of care treatment alone using quality of life questionnaires (EPIC-26).
Patient-reported quality of life | 5 years
  Determine if the addition of intermittent enzalutamide to standard of care treatment results in a patient-reported quality of life difference compared to standard of care treatment alone using quality of life questionnaires (FACT-P).
Patient-reported quality of life | 5 years
  Determine if the addition of intermittent enzalutamide to standard of care treatment results in a patient-reported quality of life difference compared to standard of care treatment alone using quality of life questionnaires (FACT-Fatigue).
Physician-reported toxicity | 5 years
  Determine if the addition of intermittent enzalutamide to standard of care treatment results in a physician-reported difference in acute and late toxicities compared to standard of care treatment alone assessed by CTCAE Toxicity 5.0.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Princess Margaret Cancer Center, Toronto, Ontario
  - Sunnybrook Research Institute, Toronto, Ontartio